CLINICAL TRIAL: NCT03022162
Title: Prevalence of Paclitaxel Induced CIPN-Related Pain and CIPN in Indian Patients With Breast Cancer : A Prospective Observational Study
Brief Title: Prevalence of Paclitaxel Induced CIPN-Related Pain and CIPN in Indian Patients With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, parmanand jain, Professor, Anaesthesiology, Critical Care & Pain. Head, Division of Pain., Tata Memorial Centre
Other Study IDs: 1758
Record Dates: First submitted 2017-01-10; First posted 2017-01-16 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer Female; Neuropathic Pain
Keywords: Neuropathic Pain, Paclitaxel, CIPN
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Since its introduction in the 1970s, Paclitaxel has been used as an effective anticancer agent against lung, breast, ovarian, leukopenia and liver cancer. But, Paclitaxel-induced peripheral neuropathy is the major dose-limiting side effect of paclitaxel.Paclitaxel induced peripheral neuropathy most commonly presents as

1. Pain
2. Burning,
3. Tingling ("pins and needles" feeling) or electric/shock-like pain,
4. Hyperalgesia,
5. Allodynia,
6. Increased sensitivity to cold or heat These symptoms are classically seen symmetrically in the distal extremities (glove and stocking distribution).

Most adverse effects associated with chemotherapy are ameliorated after cessation of the therapy, but CIPN may persist in the longterm, with 30 % patients having CIPN related symptoms beyond 6 months after completion of chemotherapy7.Understanding the epidemiology of neuropathic pain in breast cancer patients has high clinical and public health significance.

DETAILED DESCRIPTION:
PRIMARY AIM / OBJECTIVE:

Our study aims to observe the prevalence of CIPN-related pain in cancer breast patients who have received Paclitaxel based adjuvant chemotherapy where we define CIPN-related pain as - "possible" neuropathic pain in patients scoring more than 12 on Leeds Assessment of Neuropathic Symptoms and Signs pain scale (LANSS).

SECONDARY AIM / OBJECTIVE Since its introduction in the 1970s, Paclitaxel has been used as an effective anticancer agent against lung, breast, ovarian, leukopenia and liver cancer. But, Paclitaxel-induced peripheral neuropathy is the major dose-limiting side effect of paclitaxel.Paclitaxel induced peripheral neuropathy most commonly presents as

1. Pain
2. Burning,
3. Tingling ("pins and needles" feeling) or electric/shock-like pain,
4. Hyperalgesia,
5. Allodynia,
6. Increased sensitivity to cold or heat These symptoms are classically seen symmetrically in the distal extremities (glove and stocking distribution).

Most adverse effects associated with chemotherapy are ameliorated after cessation of the therapy, but CIPN may persist in the longterm, with 30 % patients having CIPN related symptoms beyond 6 months after completion of chemotherapy7.Understanding the epidemiology of neuropathic pain in breast cancer patients has high clinical and public health significance.

MATERIALS & METHODS:

The cohort will consist of women with early breast cancer (stages I through III) who had received Paclitaxel chemotherapy for breast cancer as per the Institutional guidelines within the preceding two years. History suggestive of pre-existing neuropathy will be noted.

1. All patients (who fulfill the inclusion criteria) visiting Tata Memorial hospital during Feb2017 2016 to June 2017 will be examined in the Medical Oncology OPD by one of the investigators and the current CIPN and CIPN-related pain score will be documented by using the NCI-CTCAE and LANSS scale. Then, the patients will be questioned for thepresence of similar neuropathic symptoms before starting, after starting and during Paclitaxel the chemotherapy and their replies will be recorded in the.
2. Patients who had received adjuvant chemotherapy with Paclitaxel but who could not complete their chemotherapy due to Paclitaxel induced adverse effects other than peripheral neuropathy for eg hypersensitivity to Paclitaxel will be screened but their data will be excluded from final data assessment.

2. Use of 1. Acetyl-L-carnitine (ALC) 2. Amifostine 3. Amitriptyline 4. CaMg 5. Diethyldithio-carbamate (DDTC) 6. Glutathione (GSH) 7. Nimodipine 8. All-trans-retinoic acid 9. rhuLIF 10. Vitamin E during Paclitaxel chemotherapy will be noted based on history and examination of charts.

For CIPN-related pain: The Leeds Assessment of Neuropathic Symptoms and Signs pain scale (LANSS) is a simple and valid 7-item tool for identifying patients whose pain is dominated by neuropathic mechanisms. Each item is a binary response (yes or no) to the presence of symptoms (5 items) or clinical signs (2 items). If score > 12, neuropathic mechanisms are likely to be contributing to the patient's pain.

NCI-CTCAE : The National Cancer Institute - Common Terminology Criteria for Adverse Events v4.0, NCI-CTCAE most recently updated in 2010, will be used for grading CIPN. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for CIPN. Paclitaxel induced CIPN is defined as NCI-CTCAE Grade 2 or above.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed Primary breast cancer
2. Patients who had received adjuvant chemotherapy with Paclitaxel and who have completed their Paclitaxel chemotherapy within the preceding 2 years i.e. between 1stAugust 2014 to 31st July 2016.

Exclusion Criteria:

1. Age below 18 years
2. On current Paclitaxel chemotherapy
3. Patients with radiological evidence of bone metastases.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort will consist of all female patients with primary breast cancer who received adjuvant Paclitaxel chemotherapy within the preceding 2 year period, visiting TMH from December 2017 to May 2018.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of Paclitaxel induced CIPN-related pain | 2 years post Paclitaxel Chemotherapy
  CIPN-related pain is defined as - neuropathic pain as a result of chemotherapy induced nerve damage .
  All patients (who fulfill the inclusion criteria) visiting Tata Memorial Hospital during Feb2017 to Jun2017will be examined in the Medical Oncology OPD by one of the investigators and the current CIPN-related pain score will be documented by using the LANSS scale.
  LANSS score>12 will be considered as possible CIPN-related pain for statistical analysis

SECONDARY OUTCOMES:
Prevalence of Paclitaxel induced CIPN | 2 years post Paclitaxel Chemotherapy
  CIPN defined as - neuropathy symptoms (other than pain) as a result of chemotherapy induced nerve damage .
  All patients (who fulfill the inclusion criteria) visiting Tata Memorial Hospital during Feb2017 to Jun2017will be examined in the Medical Oncology OPD by one of the investigators and the current CIPN score will be documented by using the NCI-CTCAE v4.0 grading.
  Paclitaxel induced CIPN is defined as NCI-CTCAE Grade 2 or above for statistical analysis
temporal characteristics and risk factors of CIPN-related pain | 2 years post Paclitaxel Chemotherapy
  The distribution, appearance and disappearance of syptoms related to CIPN will be based on special questionnaire.
Use of Agents offered with an intend to prevent CIPN | 2 years post Paclitaxel Chemotherapy
  Use of 1. Acetyl-L-carnitine (ALC) 2. Amifostine 3. Amitriptyline 4. CaMg 5. Diethyldithio-carbamate (DDTC) 6. Glutathione (GSH) 7. Nimodipine 8. All-trans-retinoic acid 9. rhuLIF 10. Vitamin E during Paclitaxel chemotherapy will be noted based on history and examination of charts

CONTACTS AND LOCATIONS:
Overall Officials: Anuja Bidkar, DNBAnes, Study Chair — Tata Memorial Centre; Aparna Chatterjee, MDAnes, Study Chair — Tata Memorial Centre; Sudeep Gupta, DMOnco, Study Chair — Tata Memorial Centre; Parmanand Jain, MDAnes, Principal Investigator — Tata Memorial Centre
Locations (1):
- Anuja Bidkar, Thane, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hough SW, Kanner RM. "Cancer Pain Syndromes" in Principles & Practice of Pain Medicine edited by Warfield, Carol A.; Bajwa, Zahid H. , 2nd Edition (McGraw-Hill, 2004) p 456.
- [Result] Treede RD, Jensen TS, Campbell JN, Cruccu G, Dostrovsky JO, Griffin JW, Hansson P, Hughes R, Nurmikko T, Serra J. Neuropathic pain: redefinition and a grading system for clinical and research purposes. Neurology. 2008 Apr 29;70(18):1630-5. doi: 10.1212/01.wnl.0000282763.29778.59. Epub 2007 Nov 14. PMID 18003941
- [Result] Grond S, Radbruch L, Meuser T, Sabatowski R, Loick G, Lehmann KA. Assessment and treatment of neuropathic cancer pain following WHO guidelines. Pain. 1999 Jan;79(1):15-20. doi: 10.1016/S0304-3959(98)00138-9. PMID 9928771
- [Result] Wolf S, Barton D, Kottschade L, Grothey A, Loprinzi C. Chemotherapy-induced peripheral neuropathy: prevention and treatment strategies. Eur J Cancer. 2008 Jul;44(11):1507-15. doi: 10.1016/j.ejca.2008.04.018. Epub 2008 Jun 18. PMID 18571399
- [Result] Smith BH, Lee J, Price C, Baranowski AP. Neuropathic pain: a pathway for care developed by the British Pain Society. Br J Anaesth. 2013 Jul;111(1):73-9. doi: 10.1093/bja/aet206. PMID 23794648
- [Result] Ventzel L, Jensen AB, Jensen AR, Jensen TS, Finnerup NB. Chemotherapy-induced pain and neuropathy: a prospective study in patients treated with adjuvant oxaliplatin or docetaxel. Pain. 2016 Mar;157(3):560-568. doi: 10.1097/j.pain.0000000000000404. PMID 26529271
- [Result] Seretny M, Currie GL, Sena ES, Ramnarine S, Grant R, MacLeod MR, Colvin LA, Fallon M. Incidence, prevalence, and predictors of chemotherapy-induced peripheral neuropathy: A systematic review and meta-analysis. Pain. 2014 Dec;155(12):2461-2470. doi: 10.1016/j.pain.2014.09.020. Epub 2014 Sep 23. PMID 25261162
- [Result] Jensen TS, Baron R, Haanpaa M, Kalso E, Loeser JD, Rice ASC, Treede RD. A new definition of neuropathic pain. Pain. 2011 Oct;152(10):2204-2205. doi: 10.1016/j.pain.2011.06.017. Epub 2011 Jul 18. No abstract available. PMID 21764514
- [Result] Finnerup NB, Haroutounian S, Kamerman P, Baron R, Bennett DLH, Bouhassira D, Cruccu G, Freeman R, Hansson P, Nurmikko T, Raja SN, Rice ASC, Serra J, Smith BH, Treede RD, Jensen TS. Neuropathic pain: an updated grading system for research and clinical practice. Pain. 2016 Aug;157(8):1599-1606. doi: 10.1097/j.pain.0000000000000492. PMID 27115670